CLINICAL TRIAL: NCT04282447
Title: Screening of NASH in Oupatients Followed in Various Hospital Specialty Clinics at the University Hospital of Strasbourg
Acronym: NASH-SPE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7376
Record Dates: First submitted 2020-02-21; First posted 2020-02-24 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-02

CONDITIONS: Nonalcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the present study is to assess, by using a simple algorithm combining FIB-4 and Fibroscan, the prevalence of NASH with advanced fibrosis in outpatients followed in various hospital specialty clinics other than hepato/gastroenterology and to examine risk factors associated with this condition. The prevalence of NASH will be investigated among 6 cohorts of outpatients followed in different hospital specialty clinics at Hôpitaux Universitaires de Strasbourg.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* outpatients followed at specialty clinics in HUS and at risk of NAFLD: with at least one metabolic risk factor (overweight, diabetes mellitus, hypertension, hypertriglyceridemia) and/or elevated transaminases and/or liver steatosis on US.
* endocrinology cohort : type 2 diabetes patients
* infectious disease cohort : HIV positive patients
* rheumatology cohort : patients with psoriasis, gout or rheumatoid arthritis
* nephrology cohort : patients with chronic kidney disease such as diabetic nephropathy or hypertensive nephropathy, including those receiving hemodialysis.
* cardiology cohorts: patients with history of angina, myocardial infarction, stroke or arteritis of lower limbs.
* internal medicine cohort: patients with auto immune systemic diseases such as lupus, sclerosis or rheumatoid arthritis.
* subjects who have given their informed consent
* Subjects affiliated to a social security system

Exclusion Criteria:

* alcohol consumption > 30g/d in male or > 20g/d in female in the past 6 months
* history of chronic viral hepatitis
* history of liver auto immune disease, genetic hemochromatosis, Wilson disease
* biliary disease, bile duct obstruction
* drug-induced liver injury
* secondary liver cancer or other active cancer
* organ graft
* use of medications associated with secondary NAFLD (corticosteroids, tamoxifen, amiodarone, methotrexate).
* congestive heart failure
* AIDS
* pregnancy, breastfeeding
* no information could be given to the patient (subject faces emergency situation, comprehension difficulties, etc.)
* patient under guardianship
* patients under judicial protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients followed at specialty clinics in HUS and at risk of NAFLD: with at least one metabolic risk factor (overweight, diabetes mellitus, hypertension, hypertriglyceridemia) and/or elevated transaminases and/or liver steatosis on US.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-08-14 (Actual); Primary Completion 2020-08-14 (Actual); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Estimated prevalence of NASH with advanced fibrosis among several hospital specialty clinics | 3 months
  To assess the estimated prevalence of NASH , calcul of the FIB4

CONTACTS AND LOCATIONS:
Locations (1):
- Les Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided